CLINICAL TRIAL: NCT03824821
Title: Assessing Associations Between IBS Symptoms, Nutrition and QoL in IBS Patients Using a Questionnaire
Acronym: IBSQUtrition
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government); Ingredia S.A. (Industry); Nexira (Industry); Naturex (Other); Bioiberica (Industry); Wecare (Other); Roquette Freres (Industry); Darling (Unknown); Winclove Probiotics B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18/06
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Nutrition; Irritable Bowel Syndrome; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBS
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study is a cross-sectional observational study design that aimed to include 2000 IBS patients. We used several validated questionnaires, to assess IBS characteristics (such as subtype, severity), psychological features (QoL, anxiety and depression) and assess nutritional triggers.

Subjects filled in the questionnaire online, and was spread across the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* IBS-like symptoms

Exclusion Criteria:

* younger than 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: There were no strict inclusion and exclusion criteria, since many IBS patients do not have an official diagnosis of IBS. therefore, the ROME IV diagnostic criteria were included in the questionnaire, to assess whether subjects fit within the IBS profile.
Sampling Method: Probability Sample
Enrollment: 2076 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
IBS subtype | 1 day (once )
  Assessed using the Validated Bristol stool chart
IBS severity | 1 day (once )
  Assessed by the validated Symptom severity scale (IBS-SSS), rangeing from 0 - 500; 0 very low and 500 very severe case
Nutrition questionnaire | 1 day (once )
  We composed a questionnaire containing 44 identified nutritional triggers from literature, and asked subjects if they had (0, no complaints), 1 little complaints, 2 severe complaints, after eating that product.
Birmingham symptom questionnaire | 1 day (once )
  Validated questionnaire that assesses symptoms for three domains: pain, diarrhoea and constipation

SECONDARY OUTCOMES:
Irritable bowel syndrome Quality of Life questionnaire | 1 day (once )
  We used the validated IBS-QOL which asked 44 questions about quality of life related to IBS. Score ranged from 0 - 100: 100 indicating a very high quality of life, 0 indicating a very poor quality of life
Hospital Anxiety and Depression Score (HADS) | 1 day (once )
  We used the validated HADS questionnaire to assess anxiety and depression in IBS patients. This questionnaire gives 2 scores: one for anxiety and depression. Scores range from 0-21, a score above 8 can be referred to as being a case for having anxiety or depression
treatment options currently used | 1 day (once )
  We self-composed a questionnaire to assess what type of treatments patients already used, and what their perceived effect was.
Rome IV criteria | 1 day (once )
  Validated questions to check whether a subject fits within the profile of IBS

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided